CLINICAL TRIAL: NCT01098240
Title: A RANDOMIZED PHASE 2A, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY OF THE EFFICACY AND SAFETY OF CP-601,927 AUGMENTATION OF ANTIDEPRESSANT THERAPY IN MAJOR DEPRESSION
Brief Title: A Study Of The Efficacy And Safety Of CP-601,927 Augmentation Of Antidepressant Therapy In Major Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3331017
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Results first posted 2013-06-26 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Major Depressive Disorder
Keywords: Antidepressant Augmentation
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Treatment (Experimental): CP-601,927
  Interventions: Drug: CP-601,927
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CP-601,927 — CP-601,927 1-2 mg twice per day, oral 1 mg tablets, for 6 weeks.
  Arms: Active Treatment
Other: Placebo — Matching placebo tablets, taken orally, twice per day, for 6 weeks.
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to: 1) Evaluate the efficacy of CP 601,927 compared to placebo in the augmentation of antidepressant therapy (ADT) in patients with Major Depressive Disorder (MDD) using the Montgomery Asberg Depression Rating Scale (MADRS). 2) Evaluate the safety and tolerability of CP 601,927 in patients with MDD on ADT.

DETAILED DESCRIPTION:
The study was stopped at interim analysis in August 2011, as stopping criteria for futility were met. There was no statistically significant change on the primary efficacy scale in favor of the drug. There was a very small chance that any additional data could change the study overall outcome. There were no concerns regarding subject safety.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy males or females aged 18-65 (inclusive).
* Patients must have a primary current diagnosis of MDD without psychotic features.
* Patients must be receiving ongoing antidepressant therapy at the time of screening. Duration of the current episode of MDD must be at least 8 weeks prior to enrollment without adequate response to treatment.

Exclusion Criteria:

* Patients with other psychiatric disorders.
* Patients who use tobacco products.
* Alcohol or substance abuse or dependence.
* Treatment with a monoamine oxidase inhibitor within 10 weeks of enrollment.
* Pregnancy or breastfeeding.
* Clinically significant abnormalities on laboratory tests, electrocardiogram, or physical or neurologic examination.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2010-06-14 (Actual); Primary Completion 2011-09-12 (Actual); Study Completion 2011-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (57):
- United States (57):
  - Arkansas Psychiatric Clinic Clinical Research Trials, P.A., Little Rock, Arkansas
  - Southwestern Research Incorporated, Beverly Hills, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Synergy Clinical Research Center, National City, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Radiant Research, Inc., Denver, Colorado
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - William B. Backus Hospital Satellite Blood Draw, Norwich, Connecticut
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Comprehensive NeuroScience, Inc., St. Petersburg, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Atlanta Institute of Medicine and Research, Atlanta, Georgia
  - AMR-Baber Research Inc., Naperville, Illinois
  - Psychiatric Medicine Associates, LLC., Skokie, Illinois
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - Clinco, Terre Haute, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - Louisiana Clinical Research, LLC, Shreveport, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - AccelRx Research, Fall River, Massachusetts
  - Detroit Bio-Medical Laboratories, Inc., Rochester Hills, Michigan
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Social Psychiatry Research Institute, Brooklyn, New York
  - Erie County Medical Center / State University of New York at Buffalo affiliate, Buffalo, New York
  - Comprehensive NeuroScience, Inc., Fresh Meadows, New York
  - Montefiore Medical Center, The Bronx, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - Kettlie Joseph Daniels, MD, Inc., Toledo, Ohio
  - Neurology and Neuroscience Center of Ohio, Toledo, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Summit Research Network (Oregon), Inc., Portland, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - City Line Family Medicine, Bala-Cynwyd, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - University of Pennsylvania / Department of Psychiatry, Philadelphia, Pennsylvania
  - Frankford Avenue Family Practice, PC, Philadelphia, Pennsylvania
  - Lincoln Research, Lincoln, Rhode Island
  - Carolina Clinical Research Service LLC, Columbia, South Carolina
  - FutureSearch Trials, Austin, Texas
  - FutureSearch Trials of Dallas, L.P., Dallas, Texas
  - University of Texas (UT) Southwestern Medical Center at Dallas, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Radiant Research, Inc, Salt Lake City, Utah
  - University of Utah School of Medicine Department of Psychiatry Mood Disorders Clinic, Salt Lake City, Utah
  - University of Virginia Health System / Department of Psychiatry and Neurobehavioral Sciences, Charlottesville, Virginia
  - Mcguire Hall Annex, Richmond, Virginia
  - Nelson Clinic, Richmond, Virginia
  - Virginia Commonwealth University (VCU) Medical Center, Richmond, Virginia
  - Northbrooke Research Center, Brown Deer, Wisconsin
  - Dean Foundation for Health, Research and Education, Middleton, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Fava M, Ramey T, Pickering E, Kinrys G, Boyer S, Altstiel L. A randomized, double-blind, placebo-controlled phase 2 study of the augmentation of a nicotinic acetylcholine receptor partial agonist in depression: is there a relationship to leptin levels? J Clin Psychopharmacol. 2015 Feb;35(1):51-6. doi: 10.1097/JCP.0000000000000245. PMID 25422883
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3331017&StudyName=A%20Study%20Of%20The%20Efficacy%20And%20Safety%20Of%20CP-601%2C927%20Augmentation%20Of%20Antidepressant%20Therapy%20In%20Major%20Depression%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-Label Antidepressant Treatment (ADT): Participants treated with 1 of 5 allowed antidepressant agents in accordance with current product labeling, targeting the following doses by the end of week 2: escitalopram (Lexapro) (10-20 milligram/day [mg/d]), citalopram (Celexa) (20-40 mg/d), fluoxetine (Prozac, Sarafem) (20-60 mg/d), paroxetine controlled-release (CR) (Paxil CR) (37.5-62.5 mg/d), sertraline (Zoloft) (100-200 mg/d), for up to 8 weeks in open-label phase.
- CP-601,927 + ADT: Participants treated with CP-601,927 1 mg every evening (QPM) for 3 days, then 1 mg twice daily (BID) for 3 days, then 2 mg BID on Day 7 of dosing in the double-blind phase. Dose in participants experiencing intolerable nausea may be reduced to 1 mg BID for 6 weeks and a 7-10 day follow-up period. Background ADT (continued from Open-Label ADT) was applied in the double-blind phase.
- Placebo + ADT: Placebo matched to CP-601,927 1 mg QPM for 3 days, then CP-601,927 1 mg BID for 3 days, and then CP-601,927 2 mg BID on Day 7 of dosing in the double-blind phase. Dose in participants experiencing intolerable nausea may be reduced to 1 mg BID for 6 weeks and a 7-10 day follow-up period. Background ADT (continued from Open-Label ADT) was applied in the double-blind phase.
Period: Open-Label Phase
Arm/Group | Open-Label Antidepressant Treatment (ADT) | CP-601,927 + ADT | Placebo + ADT
Started | 297 | 0 | 0
Completed | 162 | 0 | 0
Not Completed | 135 | 0 | 0
Not completed — Study Terminated by Sponsor | 27 | 0 | 0
Not completed — Protocol Violation | 4 | 0 | 0
Not completed — Lost to Follow-up | 13 | 0 | 0
Not completed — Other | 19 | 0 | 0
Not completed — Did Not Meet Entrance Criteria | 50 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0
Not completed — Adverse Event | 12 | 0 | 0
Period: Double-Blind Phase
Arm/Group | Open-Label Antidepressant Treatment (ADT) | CP-601,927 + ADT | Placebo + ADT
Started | 0 | 77 | 85
Completed | 0 | 60 | 63
Not Completed | 0 | 17 | 22
Not completed — Study Terminated by Sponsor | 0 | 5 | 8
Not completed — Protocol Violation | 0 | 2 | 4
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Other | 0 | 2 | 2
Not completed — Did Not Meet Entrance Criteria | 0 | 1 | 0
Not completed — Insufficient Clinical Response | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 3
Not completed — Adverse Event | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Open-Label ADT: Participants treated with 1 of 5 allowed antidepressant agents in accordance with current product labeling, targeting the following doses by the end of week 2: escitalopram (Lexapro) (10-20 mg/d), citalopram (Celexa) (20-40 mg/d), fluoxetine (Prozac, Sarafem) (20-60 mg/d), paroxetine CR (Paxil CR) (37.5-62.5 mg/d), sertraline (Zoloft) (100-200 mg/d), for up to 8 weeks in open-label phase.
Arm/Group | Open-Label ADT
Number analyzed (Participants) | 297
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 113
  45 to 64 years | 181
  Greater than or equal to (>=) 65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220
  Male | 77

OUTCOME MEASURES:

1. Primary Outcome: Change From Double-blind Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) - Total Score at Week 14
Description: MADRS measures the overall severity of depressive symptoms. The MADRS had a 10-item checklist. Items are rated on a scale of 0-6, for a total numeric range of scores from 0 (depressive symptoms absent) to 60 (numerically highest level of depressive symptoms).
Time Frame: Week 8 (double-blind baseline ) and week 14 (week 6 of double-blind phase)
Population: The full analysis set, which was defined as the set of all participants who consumed at least one dose of randomized study medication, was applied for the analysis. Number Analyzed = number of participants with evaluable data at each timeframe.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- CP-601,927 + ADT: Participants treated with CP-601,927 1 mg QPM for 3 days, then 1 mg BID for 3 days, then 2 mg BID on Day 7 of dosing in the double-blind phase. Dose in participants experiencing intolerable nausea may be reduced to 1 mg BID for 6 weeks and a 7-10 day follow-up period. Background ADT (continued from Open-Label ADT) was applied in the double-blind phase.
Arm/Group | CP-601,927 + ADT | Placebo + ADT
Number analyzed (Participants) | 77 | 85
Units on a scale
  Week 8 (double-blind baseline) | 29.5 (6.00) | 29.1 (5.54)
  Change at week 14: number analyzed (Participants) | 62 | 63
  Change at week 14 | -10.3 (8.60) | -8.8 (10.40)

2. Secondary Outcome: Change From Double-blind Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) - Total Score at Weeks 9 Through 13
Description: as for outcome 1
Time Frame: Week 8 (double-blind baseline) and weeks 9 through 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-601,927 + ADT | Placebo + ADT
Number analyzed (Participants) | 77 | 85
Units on a scale
  Week 8 (double-blind baseline) | 29.5 (6.00) | 29.1 (5.54)
  Change at Week 9: number analyzed (Participants) | 76 | 82
  Change at Week 9 | -2.4 (4.68) | -3.3 (5.35)
  Change at Week 10: number analyzed (Participants) | 71 | 80
  Change at Week 10 | -4.7 (6.65) | -4.6 (6.85)
  Change at Week 11: number analyzed (Participants) | 67 | 71
  Change at Week 11 | -7.0 (7.78) | -6.0 (8.06)
  Change at Week 12: number analyzed (Participants) | 64 | 73
  Change at Week 12 | -8.5 (8.08) | -7.4 (8.83)
  Change at week 13: number analyzed (Participants) | 65 | 68
  Change at week 13 | -8.6 (8.16) | -7.9 (9.37)

3. Secondary Outcome: Change From Double-blind Baseline in Hamilton Depression Scale 25-item (HAM-D25) - Total Score at Weeks 9 Through 14
Description: The HAM-D25 is the 25-item version of a scale used to assess the range of depressive symptoms including depressed mood, work and activities, sleep, suicidal thinking, psychomotor agitation/retardation, appetite, sexual interest, anxiety, somatic symptoms, and cognitive symptoms. The items on the HAM-D were rated on a scale of 0-2 or 0-4, for a total numeric range of scores from 0 (depressive symptoms absent) to 72 (numerically highest level of depressive symptoms).
Time Frame: Weeks 8 (double-blind baseline) through 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-601,927 + ADT | Placebo + ADT
Number analyzed (Participants) | 77 | 85
Units on a scale
  Week 8 (double-blind baseline) | 26.4 (4.25) | 26.3 (4.96)
  Change at week 9: number analyzed (Participants) | 76 | 82
  Change at week 9 | -3.0 (4.49) | -3.0 (5.25)
  Change at week 10: number analyzed (Participants) | 71 | 80
  Change at week 10 | -4.4 (6.57) | -4.7 (5.78)
  Change at week 11: number analyzed (Participants) | 67 | 71
  Change at week 11 | -5.9 (7.40) | -6.4 (7.06)
  Change at week 12: number analyzed (Participants) | 64 | 73
  Change at week 12 | -7.6 (7.63) | -6.7 (7.67)
  Change at week 13: number analyzed (Participants) | 65 | 68
  Change at week 13 | -8.0 (7.22) | -7.3 (7.90)
  Change at week 14: number analyzed (Participants) | 62 | 63
  Change at week 14 | -9.1 (7.76) | -8.4 (8.99)

4. Secondary Outcome: Change From Double-blind Baseline in Bech Melancholia Subscale Score at Weeks 9 Through 14
Description: The Bech Melancholia is sum of scores on 6 items (items 1, 2, 7, 8, 10 and 13) pertaining to melancholia within HAM-D. The items are rated on a scale of 0-4, higher scores reflecting greater severity. Total possible score is 0-24.
Time Frame: Weeks 8 (double-blind baseline) through 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-601,927 + ADT | Placebo + ADT
Number analyzed (Participants) | 77 | 85
Units on a scale
  Week 8 (double-blind baseline) | 11.6 (1.90) | 11.6 (2.05)
  Change at week 9: number analyzed (Participants) | 76 | 82
  Change at week 9 | -1.3 (2.31) | -1.5 (2.48)
  Change at week 10: number analyzed (Participants) | 71 | 80
  Change at week 10 | -2.1 (3.07) | -2.0 (2.87)
  Change at week 11: number analyzed (Participants) | 67 | 71
  Change at week 11 | -3.0 (3.55) | -2.7 (3.38)
  Change at week 12: number analyzed (Participants) | 64 | 73
  Change at week 12 | -3.6 (3.65) | -3.0 (3.40)
  Change at week 13: number analyzed (Participants) | 65 | 68
  Change at week 13 | -3.8 (3.56) | -3.2 (3.69)
  Change at week 14: number analyzed (Participants) | 62 | 63
  Change at week 14 | -4.3 (3.87) | -3.7 (4.15)

5. Secondary Outcome: Change From Double-blind Baseline in Clinical Global Impression - Severity (CGI-S) at Weeks 9, 10, 12, and 14
Description: CGI-S was defined as 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill participants). Higher score = more affected.
Time Frame: Week 8 (double-blind baseline) and weeks 9, 10, 12, 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-601,927 + ADT | Placebo + ADT
Number analyzed (Participants) | 77 | 85
Units on a scale
  Week 8 (double-blind baseline) | 4.2 (0.59) | 4.2 (0.67)
  Change at week 9: number analyzed (Participants) | 76 | 82
  Change at week 9 | -0.2 (0.49) | -0.2 (0.60)
  Change at week 10: number analyzed (Participants) | 71 | 80
  Change at week 10 | -0.5 (0.81) | -0.5 (0.83)
  Change at week 12: number analyzed (Participants) | 64 | 72
  Change at week 12 | -0.8 (1.01) | -0.7 (1.14)
  Change at week 14: number analyzed (Participants) | 62 | 63
  Change at week 14 | -1.1 (1.11) | -1.0 (1.18)

6. Secondary Outcome: Change From Double-blind Baseline in Sheehan Irritability Scale (SIS) Total Score at Weeks 11 and 14
Description: The SIS is to rate suffering with regard to irritability symptoms. The degree to which irritability interferes with work, social and family function is also queried. The total SIS score is the sum of 7 items. Each item is rated on a scale of 0-10, for a total numeric range of scores from 0 (not at all) to 70 (extremely). The SIS also records the number of days impaired by irritability.
Time Frame: Weeks 8 (double-blind baseline), 11 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-601,927 + ADT | Placebo + ADT
Number analyzed (Participants) | 77 | 85
Units on a scale
  Week 8 (double-blind baseline): number analyzed (Participants) | 77 | 84
  Week 8 (double-blind baseline) | 36.1 (13.21) | 34.8 (13.68)
  Change at week 11: number analyzed (Participants) | 66 | 71
  Change at week 11 | -9.3 (14.41) | -7.3 (13.70)
  Change at week 14: number analyzed (Participants) | 62 | 62
  Change at week 14 | -12.3 (15.80) | -10.4 (17.11)

7. Secondary Outcome: Change From Double-blind Baseline in Sheehan Disability Scale (SDS) Total Score at Weeks 11 and 14
Description: SDS is defined as a self-administered tool that measures functional impairment including work/school, social life, and family life/home responsibilities. Items are rated on a scale of 0-10 visual analog scale (0=not at all impaired, 10=extremely impaired), for a total numeric range of scores from 0 (not at all impaired) to 30 (extremely impaired).
Time Frame: Weeks 8 (double-blind baseline), 11 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-601,927 + ADT | Placebo + ADT
Number analyzed (Participants) | 77 | 85
Units on a scale
  Week 8 (double-blind baseline): number analyzed (Participants) | 61 | 68
  Week 8 (double-blind baseline) | 19.0 (5.88) | 18.5 (5.30)
  Change at week 11: number analyzed (Participants) | 45 | 52
  Change at week 11 | -5.6 (6.98) | -3.8 (6.33)
  Change at week 14: number analyzed (Participants) | 41 | 44
  Change at week 14 | -6.6 (7.98) | -5.7 (8.21)

8. Secondary Outcome: Change From Double-blind Baseline in Sheehan Disability Scale (SDS) Subscale Score at Weeks 11 and 14
Description: SDS subscale is defined as a self-administered tool that measures functional impairment in 3-item including work/school, social life, and family life/home responsibilities. Items are rated on a scale of 0-10 visual analog scale, for a total numeric range of scores from 0 (not at all impaired) to 30 (extremely impaired).
Time Frame: Weeks 8 (double-blind baseline), 11 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-601,927 + ADT | Placebo + ADT
Number analyzed (Participants) | 77 | 85
Units on a scale
  Week 8 (double-blind baseline): number analyzed (Participants) | 61 | 68
  Week 8 (double-blind baseline) | 6.0 (2.22) | 5.5 (2.66)
  Change at week 11: number analyzed (Participants) | 45 | 52
  Change at week 11 | -2.1 (2.86) | -0.9 (2.10)
  Change at week 14: number analyzed (Participants) | 41 | 44
  Change at week 14 | -2.1 (2.88) | -1.9 (2.66)

9. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Total Score at Weeks 9, 10, 12 and 14
Description: CGI-I was defined as a 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement was defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected.
Time Frame: Weeks 8 (double-blind baseline) 9, 10, 12 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-601,927 + ADT | Placebo + ADT
Number analyzed (Participants) | 77 | 85
Units on a scale
  Week 8 (double-blind baseline) | 3.7 (0.77) | 3.5 (0.66)
  Week 9: number analyzed (Participants) | 76 | 82
  Week 9 | 3.4 (0.84) | 3.2 (0.78)
  Week 10: number analyzed (Participants) | 71 | 80
  Week 10 | 3.2 (0.92) | 3.1 (0.88)
  Week 12: number analyzed (Participants) | 64 | 72
  Week 12 | 2.7 (1.05) | 2.8 (1.07)
  Week 14: number analyzed (Participants) | 62 | 63
  Week 14 | 2.5 (1.05) | 2.7 (1.03)

10. Secondary Outcome: Number of Participants With Remission at Weeks 9, 10, 12 and 14
Description: Remission was defined as response plus an absolute MADRS total score of less than or equal to 10 plus a CGI-I score less than 2 ('much' or 'very much' improved).
Time Frame: Weeks 9, 10, 12 and 14
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | CP-601,927 + ADT | Placebo + ADT
Number analyzed (Participants) | 76 | 82
Participants
  Week 9 | 1 | 0
  Week 10: number analyzed (Participants) | 71 | 80
  Week 10 | 4 | 1
  Week 12: number analyzed (Participants) | 64 | 72
  Week 12 | 5 | 9
  Week 14: number analyzed (Participants) | 62 | 63
  Week 14 | 9 | 11

11. Secondary Outcome: Number of Participants With Response at Weeks 9 Through 14
Description: Response was defined as greater than 50 percent reduction from double-blind baseline in MADRS total score.
Time Frame: Weeks 9 through 14
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | CP-601,927 + ADT | Placebo + ADT
Number analyzed (Participants) | 76 | 82
Participants
  Week 9 | 3 | 4
  Week 10: number analyzed (Participants) | 71 | 80
  Week 10 | 8 | 8
  Week 11: number analyzed (Participants) | 67 | 71
  Week 11 | 15 | 10
  Week 12: number analyzed (Participants) | 64 | 73
  Week 12 | 18 | 16
  Week 13: number analyzed (Participants) | 65 | 68
  Week 13 | 23 | 20
  Week 14: number analyzed (Participants) | 62 | 63
  Week 14 | 22 | 20

12. Secondary Outcome: Population Pharmacokinetics
Description: Population pharmacokinetic analysis involved mixed effects modeling using nonlinear mixed effects modeling (NONMEM) software. The intent of this analysis was to establish a basic population pharmacokinetic model for CP-601,927 and to determine inter-individual and residual variability in population clearance, and volume of distribution of drug. Relationship of demographic variables (gender, age, body weight, height and ethnicity), concomitant medications and measures of altered hepatic and renal function were examined by fitting measured CP-601,927 concentrations
Time Frame: Weeks 11,12 and 14
Population: Data for this outcome measure was not collected and reported because the planned analysis (data collection) was not done as the study was stopped early for futility.
Reporting Status: Not Posted

13. Secondary Outcome: Plasma CP-601,927 Concentration
Description: Blood samples were collected for plasma CP-601,927 concentration analysis which was summarized by mean and standard deviation.
Time Frame: Week 11, 12 and 14
Population: All randomized participants with at least one dose of study medication in DB (double blind) phase and one valid plasma concentration measurement collected during the DB phase was be included in the analyses of the PK endpoints. Number Analyzed = number of participants with evaluable data at each timeframe.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-601,927 + ADT
Number analyzed (Participants) | 60
ng/mL
  Week 11 at 1 Hour: number analyzed (Participants) | 53
  Week 11 at 1 Hour | 5.80 (3.42)
  Week 11 at 2 Hours: number analyzed (Participants) | 53
  Week 11 at 2 Hours | 5.90 (3.13)
  Week 12: number analyzed (Participants) | 56
  Week 12 | 6.24 (3.85)
  Week 14 at 1 Hour | 5.36 (3.83)
  Week 14 at 2 Hour: number analyzed (Participants) | 57
  Week 14 at 2 Hour | 5.39 (3.89)

14. Other Pre Specified Outcome: The Sheehan Suicidality Tracking Scale (STS)
Description: The Sheehan Suicidality Tracking Scale (STS) measures treatment-emergent suicidal ideation as well as behaviors. It can be administered by a clinician or filled in by a participant. Prior to analysis, the STS was mapped to the Columbia Classification Algorithm of Suicide Assessment(C-CASA) categories, which has 9-item including completed suicide, suicide attempt, preparatory acts, suicidal ideation, self-injurious behavior, self-injurious no intent, unknown fatal,unknown non-fatal or other not deliberate. Participants who were mapped to C-CASA items were reported.
Time Frame: Week 8 (double-blind baseline) and weeks 9 through 14
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | CP-601,927 + ADT | Placebo + ADT
Number analyzed (Participants) | 77 | 85
Participants
  Week 8: suicidal ideation | 11 | 13
  Week 8: no suicidal behavior and risk | 66 | 72
  Week 9: suicidal ideation: number analyzed (Participants) | 72 | 79
  Week 9: suicidal ideation | 10 | 8
  Week 9: self-injurious, no intent: number analyzed (Participants) | 72 | 79
  Week 9: self-injurious, no intent | 1 | 0
  Week 9: no suicidal behavior and risk: number analyzed (Participants) | 72 | 79
  Week 9: no suicidal behavior and risk | 61 | 71
  Week 10: suicidal ideation: number analyzed (Participants) | 69 | 74
  Week 10: suicidal ideation | 12 | 7
  Week 10: no suicidal behavior and risk: number analyzed (Participants) | 69 | 74
  Week 10: no suicidal behavior and risk | 57 | 67
  Week 11: suicidal ideation: number analyzed (Participants) | 64 | 71
  Week 11: suicidal ideation | 8 | 5
  Week 11: no suicidal behavior and risk: number analyzed (Participants) | 64 | 71
  Week 11: no suicidal behavior and risk | 56 | 66
  Week 12: suicidal ideation: number analyzed (Participants) | 63 | 70
  Week 12: suicidal ideation | 6 | 5
  Week 12: no suicidal behavior and risk: number analyzed (Participants) | 63 | 70
  Week 12: no suicidal behavior and risk | 57 | 65
  Week 13: suicidal ideation: number analyzed (Participants) | 62 | 63
  Week 13: suicidal ideation | 5 | 5
  Week 13: no suicidal behavior and risk: number analyzed (Participants) | 62 | 63
  Week 13: no suicidal behavior and risk | 57 | 58
  Week 14: suicidal ideation: number analyzed (Participants) | 75 | 81
  Week 14: suicidal ideation | 5 | 6
  Week 14: no suicidal behavior and risk: number analyzed (Participants) | 75 | 81
  Week 14: no suicidal behavior and risk | 70 | 75

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Open-Label ADT | CP-601,927 + ADT | Placebo + ADT
Serious Adverse Events (participants affected / at risk) | 3/297 | 1/77 | 1/85
Other Adverse Events (participants affected / at risk) | 210/297 | 58/77 | 61/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label ADT (N=297) | CP-601,927 + ADT (N=77) | Placebo + ADT (N=85)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label ADT (N=297) | CP-601,927 + ADT (N=77) | Placebo + ADT (N=85)
Palpitations (Cardiac disorders) | 4 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 2 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 5 | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 4 | 1
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 11 | 2 | 3
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 28 | 4 | 5
Dry mouth (Gastrointestinal disorders) | 17 | 4 | 8
Dyspepsia (Gastrointestinal disorders) | 6 | 3 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 7 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 2 | 0 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1 | 0
Gingival swelling (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 39 | 11 | 12
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Tongue cyst (Gastrointestinal disorders) | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 3 | 0 | 2
Vomiting (Gastrointestinal disorders) | 3 | 2 | 1
Asthenia (General disorders) | 2 | 1 | 1
Chills (General disorders) | 1 | 0 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 18 | 3 | 13
Feeling abnormal (General disorders) | 0 | 1 | 0
Feeling hot (General disorders) | 1 | 0 | 1
Feeling jittery (General disorders) | 3 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
Irritability (General disorders) | 12 | 2 | 5
Local swelling (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 4 | 1 | 0
Pain (General disorders) | 2 | 1 | 0
Pyrexia (General disorders) | 4 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0
Multiple allergies (Immune system disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 1
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0
Conjunctivitis infective (Infections and infestations) | 1 | 0 | 1
Fungal infection (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 1 | 0
Gingival infection (Infections and infestations) | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 6 | 1 | 2
Laryngitis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 10 | 2 | 2
Oral infection (Infections and infestations) | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 5 | 1 | 2
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 24 | 6 | 4
Urinary tract infection (Infections and infestations) | 6 | 4 | 2
Viral infection (Infections and infestations) | 1 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 3 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1
Blood glucose decreased (Investigations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 2 | 1 | 3
Colonoscopy (Investigations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 1
Positive Rombergism (Investigations) | 0 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 2 | 0
Weight increased (Investigations) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Food craving (Metabolism and nutrition disorders) | 2 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 4 | 1 | 3
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Akathisia (Nervous system disorders) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 22 | 5 | 4
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 42 | 16 | 12
Hypersomnia (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0
Lethargy (Nervous system disorders) | 2 | 1 | 1
Memory impairment (Nervous system disorders) | 2 | 0 | 1
Migraine (Nervous system disorders) | 1 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Oromandibular dystonia (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 4 | 1 | 0
Poor quality sleep (Nervous system disorders) | 2 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 2 | 0 | 1
Retrograde amnesia (Nervous system disorders) | 1 | 0 | 0
Sedation (Nervous system disorders) | 6 | 1 | 1
Sinus headache (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 18 | 4 | 4
Syncope (Nervous system disorders) | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 3 | 2 | 0
Abnormal dreams (Psychiatric disorders) | 3 | 5 | 3
Affective disorder (Psychiatric disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 2 | 0 | 1
Anger (Psychiatric disorders) | 0 | 0 | 1
Anorgasmia (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 8 | 2 | 1
Apathy (Psychiatric disorders) | 2 | 0 | 1
Bruxism (Psychiatric disorders) | 3 | 0 | 1
Depression (Psychiatric disorders) | 4 | 0 | 1
Emotional disorder (Psychiatric disorders) | 1 | 0 | 1
Initial insomnia (Psychiatric disorders) | 3 | 1 | 1
Insomnia (Psychiatric disorders) | 24 | 10 | 10
Libido decreased (Psychiatric disorders) | 7 | 1 | 2
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Middle insomnia (Psychiatric disorders) | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 2 | 1 | 0
Nightmare (Psychiatric disorders) | 0 | 3 | 2
Orgasm abnormal (Psychiatric disorders) | 1 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 1
Panic reaction (Psychiatric disorders) | 0 | 1 | 0
Paranoia (Psychiatric disorders) | 2 | 0 | 0
Personality disorder (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0
Sleep terror (Psychiatric disorders) | 0 | 1 | 0
Suspiciousness (Psychiatric disorders) | 1 | 0 | 1
Tachyphrenia (Psychiatric disorders) | 0 | 1 | 0
Terminal insomnia (Psychiatric disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0
Ejaculation delayed (Reproductive system and breast disorders) | 1 | 1 | 0
Erection increased (Reproductive system and breast disorders) | 1 | 0 | 0
Menstruation delayed (Reproductive system and breast disorders) | 0 | 0 | 1
Polycystic ovaries (Reproductive system and breast disorders) | 0 | 1 | 0
Polymenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Yawning (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Colon polypectomy (Surgical and medical procedures) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 4 | 0 | 1
Hypertension (Vascular disorders) | 2 | 3 | 0
Hypotension (Vascular disorders) | 2 | 2 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.